CLINICAL TRIAL: NCT02271243
Title: Using Microbial Genomics to Elucidate the Source of Central-line Associated Bloodstream Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Priebe, Staff Physician Critical Care & Infectious Disease, Boston Children's Hospital
Other Study IDs: P00012105
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Laboratory-confirmed Bloodstream Infection; Central Line-associated Bloodstream Infections; Mucosal Barrier Injury
Keywords: Central line-associated bloodstream infections; mucosal barrier injury; laboratory-confirmed bloodstream infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacteria growing from swab of oral cavity, sputum, skin, stool, and blood; stool and plasma samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subject with suspected MBI
- Subjects without suspected MBI

SUMMARY:
Central line-associated bloodstream infections (CLABSIs) are the most common healthcare-associated infection in children and are associated with morbidity and mortality. This study will attempt to identify the source of bloodstream infections (BSIs) in children with CLABSI because we hypothesize that many of the BSIs that are currently classified as CLABSIs are actually laboratory-confirmed bloodstream infections (LCBI) that may be a result of mucosal barrier injury (MBI), also known as MBI-LCBI. In order to study this, we will isolate bacteria from multiple body sites of children that have BSI in order to compare these bacteria to the strain growing in their blood using whole-genome DNA sequencing. We will also evaluate biomarkers of MBI of the respiratory tract and GI tract.

DETAILED DESCRIPTION:
This is a prospective cohort pilot study at Boston Children's Hospital (BCH) that will explore the source of presumed CLABSI, which we believe may actually have multiple possible sources including MBI. We plan to enroll all inpatient children at BCH who meet the Centers for Disease Control and Prevention (CDC) definition of MBI-LCBI as well as children who meet the criteria for CLABSI without MBI. For all enrolled patients, we will collect samples from the oral cavity, respiratory tract, skin, and stool. These samples will be cultured in order to see if the same microbial species and strain(s) growing from the blood also grow from these other sites. Cultures will then have isolated colonies selected for whole-genome DNA sequencing to allow assessment of genomic diversity between body sites. Stool and blood samples will be tested for markers of MBI. All patient enrollment and sample collection will be done at BCH.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Boston Children's Hospital
* Central venous catheter of any type including peripherally inserted central catheters (PICC) in any location.
* Laboratory-confirmed bloodstream infection (LCBI) diagnosed by a clinical blood culture growing certain Gram-negative rods

Exclusion Criteria:

* Patients with CDC-defined secondary bloodstream infections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with CLABSI
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phylogenetic relationships (on SNP scale) of bacteria isolated from different body sites | Up to 2 years
  Phylogeny will be determined using whole-genome DNA sequences of multiple bacterial colonies that grow from each body site.

SECONDARY OUTCOMES:
Levels of biomarkers of MBI in the blood and stool (citrulline in blood, calprotectin in stool) | Up to 2 years
  Low citrulline and high calprotectin indicate GI tract mucosal barrier injury.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Priebe, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States